CLINICAL TRIAL: NCT04884399
Title: A Randomized, Double-blind, Two-group Parallel, Positive-controlled Clinical Phase I Trial Comparing the Safety, Pharmacokinetics, Pharmacodynamics and Efficacy of CMAB818 and Lucentis® in Patients With Wet Age-related Macular Degeneration.
Brief Title: Phase I Study to Compare CMAB818 Injection and Lucentis® in Patients With Wet AMD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Biomabs Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMAB818-I-001
Record Dates: First submitted 2021-05-06; First posted 2021-05-13 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Wet Age-related Macular Degeneration
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMAB818 (Experimental): 0.5 mg by intravitreal injection once on the first day.
  Interventions: Drug: CMAB818
- Lucentis® (Active Comparator): 0.5 mg by intravitreal injection once on the first day.
  Interventions: Drug: Lucentis®

INTERVENTIONS:
Drug: CMAB818 — vascular endothelial growth factor (VEGF) inhibitor
  Other Names: Ranibizumab Injection
  Arms: CMAB818
Drug: Lucentis® — vascular endothelial growth factor (VEGF) inhibitor
  Other Names: Ranibizumab Injection
  Arms: Lucentis®

SUMMARY:
This is a randomized, double-blind, two-group parallel, positive-controlled clinical Phase I trial comparing the safety, pharmacokinetics, pharmacodynamics and efficacy of CMAB818 and Lucentis® in patients with wet age-related macular degeneration.

DETAILED DESCRIPTION:
This is a phase I, randomized, double-blind, two-group parallel, positive-controlled clinical trial at four sites. Subjects will be sequentially enrolled according to the protocol in one of two cohorts and receive a single 0.5mg of CMAB818 or Lucentis® through intravitreal injection.

The primary objective is to assess the initial clinical safety of intravitreal injection of CMAB818 or Lucentis® in patients with wet age-related macular degeneration (wet-AMD).

The secondary objective are to assess immnogenicity, pharmacokinetic, pharmacodynamics and the initial clinical efficacy of intravitreal injection of CMAB818 or Lucentis® in patients with wet age-related macular degeneration (wet-AMD).

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent, and able to receive follow-up according to the time stipulated by the trial;
2. 50 years≤age≤80 years, male or female;
3. The target eye must meet the following requirements: newly occurring or relapsed subfoveal and perifoveal active choroidal neovascularization (CNV) lesions secondary to AMD; the best corrected visual acuity between 78-19 letters (including the boundary value, using Early Treatment of Diabetic Retinopathy Study (ETDRS) charts, equivalent to Snellen visual acuity of 20/32 to 20/400); no refractive media opacity or myosis affecting fundus examination;
4. The best corrected visual acuity of the subject's non-target eye≥19 letters (using ETDRS charts, equivalent to Snellen visual acuity of 20/400).

Exclusion Criteria:

1. Previously received anti-VEGF drug treatment in either eye within 3 months before screening (e.g., aflibercept<Eylea®>, ranibizumab<Lucentis®>, bevacizumab<Avastin®>, Conbercept<Lumitin®>, etc.);
2. Active eye infection in either eye within 1 months before screening (including but not limited to Blepharitis, Conjunctivitis infective, Keratitis, Scleritis, Endophthalmitis);
3. History of vitreous hemorrhage within 3 months before screening;
4. History or presence of uncontrolled glaucoma (defined as intraocular pressure(IOP)>25 mmHg despite treatment with maximal medical therapy),or the optic fovea/optical disc ratio of the target eye caused by severe glaucoma > 0.8;
5. Previously received subconjunctival/intravitreal corticosteroids injection within 3 months (including subconjunctival/intravitreal long-acting implants within 6 months), or local ocular corticosteroids treatment in the target eye within 1 month before screening;
6. Previously received the following ophthalmic surgery such as verteporfin photodynamic therapy (PDT), macular translocation, glaucoma filtering, subfoveal laser photocoagulation, vitrectomy and transpupillary thermotherapy, and other submacular surgery or surgery used to treat age-related macular degeneration in the target eye;
7. Other ocular diseases other than wAMD that affect the central vision, such as dry AMD, venous occlusion, uveitis, diabetic retinopathy, vascular-like streaks, pathological myopia, retinal detachment, macular hole, etc. in the target eye;
8. Aphakia (excluding intraocular lenses) or rupture of the posterior lens capsule in the target eye [except for yttrium aluminum garnet (YAG) laser posterior capsulotomy after intraocular lens implantation];
9. History of rhegmatogenous retinal detachment or macular hole retinal detachment (stage 3 or 4), with retinal detachment, retinal pigment epithelial tear, or retinal traction in the macular area and epiretinal disease in the macular area in the target eye;
10. Current use or may need to use systemic drugs that can cause crystal toxicity, such as psoralen, risedronate sodium, tamoxifen, etc.;
11. Allergy to fluorescein sodium or indocyanine green, protein products for treatment or diagnosis, and more than 2 drugs and/or non-drugs;
12. History of surgical operations (except for minimally invasive surgery that has healed) or currently unhealed wounds, moderate to severe ulcers, fractures, etc. within 1 month before screening;
13. Presence of infectious diseases that require oral, intramuscular or intravenous administration;
14. Presence of active diffuse intravascular coagulation or obvious bleeding tendency or abnormal coagulation function before screening (prothrombin time ≥ 3 seconds of upper limit of normal value, activated partial thromboplastin time ≥ 10 seconds of upper limit of normal value);
15. History of myocardial infarction, cerebral infarction, unstable angina, coronary revascularization, New York College of Cardiology (NYHA) grade ≥ grade II cardiac insufficiency, severely unstable ventricular arrhythmia, and cerebrovascular accident (including transient ischemic attack) before screening;
16. Presence of systemic immune diseases (including but not limited to systemic lupus erythematosus, immune hemolytic anemia, hyperthyroidism);
17. Uncontrolled hypertension(defined assystolic blood pressure≥160 mmHg and/or diastolic blood pressure≥100 mmHg diastolic despite treatment with antihypertensive drugs;
18. Diabetes with uncontrolled blood glucose (defined as fasting blood glucose≥7.0 mmol/L);
19. Any uncontrollable clinical problems (including but not limited to serious mental, neurological, respiratory and other system diseases, as well as malignant tumors);
20. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) higher than 1.5 times the laboratory upper limit of normal (ULN) and/or blood creatinine is higher than ULN and the investigator judges that the abnormality has clinical significance;
21. Concurrent with hepatitis B (positive hepatitis B virus surface antigen), hepatitis C (positive hepatitis C virus antibody), AIDS (positive human immunodeficiency virus antibody) or syphilis (positive syphilis antibody);
22. Pregnant and lactating women;
23. Refuse to take effective contraceptive measures during childbearing age throughout the study period;
24. Participated in any drug (excluding vitamins and minerals) and medical device clinical trials within 3 months before screening (if the drug has a long half-life and its 5 half-life time is greater than 3 months, then choose the 5 half-life time);
25. Any other situations that investigator thinks the subject is inappropriate to participate in this study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events That Are Related to Treatment | 0~42 days
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial participant graded according to the common terminology criteria for adverse events (CTCAE) v.5.0 criteria, including clinically-significant changes in physical examinations, laboratory safety tests, ECG and vital signs

SECONDARY OUTCOMES:
Number of Participants With anti-drug antibody | 0~42 days
  Blood samples were collected at the following time point: pre-dose, D14, D28, and D42
Percentage of neutralizing antibody | 0~42 days
  Subjects with a positive antibody response to ranibizumab were determined to test neutralizing antibody
AUC(0-t) | 0~42 days
  Blood samples were collected to measure the area under the concentration time curve from time 0 to last time
Cmax | 0~42 days
  Blood samples were collected to measure maximum concentration
CL | 0~42 days
  Blood samples were collected to measure clearance rate
Half-life (t1/2) | 0~42 days
  Blood samples were collected to measure half-life time
Pharmacodynamics | 0~42 days
  The plasma VEGF concentration from baseline were measured
Mean change in best corrected visual acuity (BCVA) from baseline | 0~42 days
  BCVA was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) visualacuity (VA) chart starting at a test distance of 4 meters. The BCVA score is the number of letters read correctly by the patient
Mean change in central retinal thickness from baseline | 0~42 days
  Central retinal thickness was measured using the Optical Coherence Tomography
Mean change in lesion area from baseline | 0~42 days
  The lesion area was measured using Fundus Fluorescein Angiography
Mean change in leakage area from baseline | 0~42 days
  The leakage area was measured using Fundus Fluorescein Angiography

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Wei, PhD, Study Chair — Beijing Tongren Hospital; Xiuli Zhao, PhD, Study Chair — Beijing Tongren Hospital
Locations (4):
- China (4):
  - Peking University People'S Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Shanghai General Hospital, Shanghai, Shanghai Municipality